CLINICAL TRIAL: NCT03983876
Title: Multi-center, Randomized, Open-Label, 2-Arm Parallel Study to Compare the Pharmacokinetics, Safety and Tolerability of AVT02 Administered Subcutaneously Via Prefilled Syringe or Autoinjector in Healthy Adult Volunteers (ALVOPAD PEN)
Brief Title: PK, Safety and Tolerability Study of AVT02 (Adalimumab) Pre-filled Syringe (PFS) vs, AVT02 Autoinjector (AI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVT02-GL-102
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Phase 1
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, 2-arm parallel study of AVT02 (Administered via a PFS either manually via an autoinjector, in healthy adult subjects. The subjects in both arms will receive the same dose of AVT02, but in two different delivery modes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVT02 100mg/mL in PFS (Experimental): Prefilled Syringe Arm
  Interventions: Drug: Adalimumab
- AVT02 100mg/mL in Autoinjector (Experimental): Autoinjector Arm
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — AVT02, a proposed similar biological product (biosimilar) of Humira which contains adalimumab . Adalimumab is a recombinant, fully human monoclonal immunoglobulin G1 (IgG1) antibody that binds specifically and with high affinity to the soluble and transmembrane forms of tumor necrosis factor (TNF)-α thereby inhibiting the binding of TNF-α with its receptor, and inhibiting TNF -α's biological function.
  Tumor necrosis factor-α is a naturally occurring cytokine that is key to normal inflammatory and immune responses. Elevated levels of TNF-α are found in the synovial fluid of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis patients and psoriasis plaques and play an important role in both the pathologic inflammation and joint destruction that are hallmarks of these inflammatory disease
  Other Names: Humira ATC code L04AB0

SUMMARY:
This study has been designed as a multicentre, randomised, open label study of AVT02 in healthy adult subjects. The study will assess the PK, safety and tolerability of AVT02 in Pre-Filled Syringe compared to AVT02 in Autoinjector Pen. Both arms will use single dose of 40mg of AVT02 (Adalimumab)

DETAILED DESCRIPTION:
This study is designed as a multi-center, randomized, open-label, 2-arm parallel study of AVT02 administered via a PFS either manually via an autoinjector, in healthy adult subjects.

A total of 204 subjects will be recruited into this study and will be randomly assigned with a ratio of 1:1 to receive either AVT02 manually or via autoinjector. As the study is open-label, both the site staff and the subjects themselves will know which treatments are being administered.

The study consists of a screening period, admission and treatment period, assessment period and end of study (EOS) visit. Subjects will undertake a screening visit between Day -28 and Day -1 to determine eligibility in the study. Those subjects that meet the eligibility criteria will be admitted to the study site on the evening prior to dosing (Day -1) when continued eligibility will be assessed.

On Day 1 prior to dosing, baseline assessments will be performed. Subjects will then be dosed according to the randomization schedule. Following dosing, PK, safety, tolerability and immunogenicity assessments will be performed according to the study schedule (Table 6). Subjects will remain confined to the study site from Day -1 to Day 3 (48 hours post-dose). Subjects will return to the study site on Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 12, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50 and Day 57.

An EOS visit will occur at study Day 64 for final study assessments. The EOS visit will also be the early termination visit if required (to be completed within 7 days of early termination wherever possible).

ELIGIBILITY:
Inclusion Criteria:To be eligible for study entry, subjects must satisfy all of the following criteria:

* Male or female healthy adult subjects willing to sign a patient information and consent form (PICF) and able to undergo protocol related procedures;
* Age: 18 to 55 years, inclusive;
* Body Mass Index: 18.5 to 32.0 kg/m2;
* No history or evidence of a clinically significant disorder, condition, or disease that, in the opinion of the investigator would pose a risk to subject safety;
* Resting supine systolic blood pressure (BP) of ≤150 mmHg and diastolic BP of ≤90 mmHg. Other vital signs showing no clinically relevant deviations according to the investigator's judgment;
* 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the investigator;
* Negative urine drug screen and negative alcohol breath test at screening and admission;
* Subjects smokes <10 cigarettes per day within 3 months of screening and is able to abide by the smoking policy of the site;
* Ability and willingness to abstain from alcohol from 48 hours prior to IP administration, during confinement in the study site until discharge from the confinement period and 24 hours prior to ambulatory visits;
* Females must have a negative pregnancy test at screening and on admission to the study site, must not be lactating and must agree to sexual abstinence or the use effective contraception, starting at screening and continue throughout the study period up to the end of study (EOS) visit;
* Male subjects and their female spouse/partners who are of childbearing potential must agree to using 2 forms of birth control (1 of which is a highly effective method and 1 must be a barrier method), or agree to sexual abstinence, starting at screening and continue throughout the study period up to the EOS visit;
* Male subject must not donate sperm starting at screening and throughout the study period up to the EOS visit;

Exclusion Criteria:To be eligible for study entry, subjects must satisfy all of the following criteria:

* Male or female healthy adult subjects willing to sign a patient information and consent form (PICF) and able to undergo protocol related procedures;
* Age: 18 to 55 years, inclusive;
* Body Mass Index: 18.5 to 32.0 kg/m2;
* No history or evidence of a clinically significant disorder, condition, or disease that, in the opinion of the investigator would pose a risk to subject safety;
* Resting supine systolic blood pressure (BP) of ≤150 mmHg and diastolic BP of ≤90 mmHg. Other vital signs showing no clinically relevant deviations according to the investigator's judgment;
* 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the investigator;
* Negative urine drug screen and negative alcohol breath test at screening and admission;
* Subjects smokes <10 cigarettes per day within 3 months of screening and is able to abide by the smoking policy of the site;
* Ability and willingness to abstain from alcohol from 48 hours prior to IP administration, during confinement in the study site until discharge from the confinement period and 24 hours prior to ambulatory visits;
* Females must have a negative pregnancy test at screening and on admission to the study site, must not be lactating and must agree to sexual abstinence or the use effective contraception, starting at screening and continue throughout the study period up to the end of study (EOS) visit;
* Male subjects and their female spouse/partners who are of childbearing potential must agree to using 2 forms of birth control (1 of which is a highly effective method and 1 must be a barrier method), or agree to sexual abstinence, starting at screening and continue throughout the study period up to the EOS visit;
* Male subject must not donate sperm starting at screening and throughout the study period up to the EOS visit;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve AUC0-t | From baseline to day 64
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUC 0-t) of AVT02 given in PFS and AVT02 given in autoinjector
Area under the plasma concentration-time curve AUC0-inf | From baseline to day 64
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUC 0-t) of AVT02 given in PFS and AVT02 given in autoinjector
Maximum serum concentration | From baseline to day 64
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUC 0-t) of AVT02 given in PFS and AVT02 given in autoinjector

SECONDARY OUTCOMES:
Pain, Tenderness, Erythema and Swelling | From baseline to day 64
  The injection sites will be monitored for pain, tenderness, erythema and swelling. Each injection site reaction will be categorised using the Injection Site Intensity Grading Scheme. All four outcome measures mentioned in the title will be measured from this one scheme. According to the Intensity Grading Scheme, the Pain, Tenderness, Erythema and Swelling will be measured as Absent (0), Mild (1), Moderate Severe(3) and Potentially Life Threatening.
Anti Drug Antibodies (ADRs) | From baseline to day 64
  Immunogenicity response will be determined from all patients treated with AVT02 from baseline to day 64 with a validated assay. Immunogenicity results (number of positive tested subjects/number of negative tested subjects; titer) will be summarized by treatment group (prefilled syringe group vs. autoinjector group). Immunogenicity assessments include antidrug antibodies (ADAs) and neutralizing antibodies (NAbs).
Adverse Events | Baseline to day 84
  Adverse events will be coded using MedDRA and grouped by system organ class and preferred term and summarised, by treatment group at the time of onset of the AE. The summary tables will present the number and percentage of total subjects and number of events, by system organ class and by preferred term. Injection related reactions will be listed and summarised by reaction using frequency counts and percentage, by treatment group

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Christchurch Clinical Studies Trust Limited, Christchurch, Chistchurch
  - Auckland Clinical Studies, Auckland

IPD SHARING:
Plan to Share IPD: No